CLINICAL TRIAL: NCT03587792
Title: Study of Binaural Squelch Effect Among Patients Undergoing Unilateral Otosclerosis Surgery: Comparison of Understanding in Noise Before-after Surgery
Brief Title: Study of Binaural Squelch Effect in Unilateral Otosclerosis
Acronym: CBOU
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.325; 2017-A02900-53 (Other: ID RCB)
Record Dates: First submitted 2018-06-04; First posted 2018-07-16 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Otosclerosis of Middle Ear; Unilateral Hearing Loss
MeSH Terms: conditions — Hearing Loss, Unilateral | interventions — Stapes Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: stapedectomy — Stapedectomy as described in literature with stapes removal, Carbon Dioxide (CO2) laser platinectomy and placement of a prothesis(piston) between the incus long process and the stapes footplate
  Other Names: platinectomy

SUMMARY:
Patients with unilateral transmission hypoacusis due to otosclerosis undergoing stapedectomy surgery will be prospectively included.

They will be undergoing a free field vocal audiometry using the Oldenburg MATRIX software to evaluated the squelch effect gain between audiometry before and after 9months after surgery.

Our hypothesis is to show a squelch effect with the rehabilitation of the binaural audition.

DETAILED DESCRIPTION:
Otosclerosis is one of the main causes of transmission hypoacusis. It can be treated with stapedectomy surgery.

But the understanding ability in noise has not been really studied. The Oldenburg MATRIX test is a well know test in audiology and allow to study the understanding in noise.

This study included all the patients coming in our center for stapedectomy for otosclerosis with controlateral audition under 30 decibels (dB) loss.

They will all undergo the MATRIX test in three situations: vocal material and noise from the front of the patient (S0N0 situation); vocal material from the front and noise from the bad-earing side (S0N-90 situation); vocal material from the front and noise from the good-earing side (S0N90 situation).

This might give three informations:

-Squelch effect which is the difference between Speech Reception Threshold (SRT) in S0N90 situation at 9month after surgery and before surgery.

The squelch effect is the ability of cortical discrimination to extract spatial cues and information providing from two different sources. So we considered the situation before surgery as a unilateral condition and the surgery rehabilitation as a bilateral condition.

* Head Shadow effect which is the difference between S0N90 and S0N-90 audiometry situations. The head shadow effect is the difference in the Speech Reception Threshold (SRT) due to diffraction effect of the physical sound wave.
* Binaural benefit which is the difference between S0N0 situation after and before surgery.

The binaural benefit is the SRT gain of both ear with same threshold comparing to a gap of threshold between the two ears.

The patients will also filled two questionnaires of quality of life: Abbreviated Profile of Hearing Aid Benefit (APHAB) and Speech and Spatial Questionnaire (SSQ).

The aim is to show the benefit of the surgery in otosclerosis for comprehension in noise.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of otosclerosis
* controlateral audiometry under 30dB loss
* the ear to be operated with a transmission over 30dB

Exclusion Criteria:

* otosclerosis which has already operated on the ear studied
* other cause of transmission hypoacusis
* transmission after surgery other 30dB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients undergoing a stapedectomy for unilateral disabled ear due to otosclerosis
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Measure of squelch effect 9 months after surgery | 9 months
  Speech reception threshold between S0N90 situation after and before surgery

SECONDARY OUTCOMES:
Measure of shadow effect 9 months after surgery | 9 months
  Comparison of Speech reception threshold between (S0N90) - (S0N-90) between 9months after surgery and before surgery
Measure of binaural benefit 9 months after surgery | 9 months
  Comparison of Speech reception threshold S0N0 between 9months after surgery and before surgery
improving quality of life : Abbreviated Profile of Hearing Aid Benefit | 9 months
  comparison of the global score and the four sub-scales: "aversiveness"; "reverberation"; "background noise"; "ease of communication" between 3 months after surgery and before surgery
Improving quality of life : Speech and Spatial Questionnaire | 9 months
  comparison of the global score and the three sub-scale: "speech hearing"; "spatial hearing"; "qualities of hearing"
Measure of squelch effect 3 months after surgery | 3 months
  Speech reception threshold between S0N90 situation after and before surgery
Measure of binaural benefit 3 months after surgery | 3 months
  Comparison of Speech reception threshold S0N0 between 3 months after surgery and before surgery
Measure of shadow effect 3 months after surgery | 3 months
  Comparison of Speech reception threshold between (S0N90) - (S0N-90) between 3 months after surgery and before surgery
improving quality of life : Abbreviated Profile of Hearing Aid Benefit | 3 months
  comparison of the global score and the four sub-scale: "aversiveness"; "reverberation"; "background noise"; "ease of communication" between 3 months after surgery and before surgery
Improving quality of life : Speech and Spatial Questionnaire | 3 months
  comparison of the global score and the three sub-scale: "speech hearing"; "spatial hearing"; "qualities of hearing" between 3 months after surgery and before surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Grenoble, Grenoble, Rhone Alpes Auvergne, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rudic M, Keogh I, Wagner R, Wilkinson E, Kiros N, Ferrary E, Sterkers O, Bozorg Grayeli A, Zarkovic K, Zarkovic N. The pathophysiology of otosclerosis: Review of current research. Hear Res. 2015 Dec;330(Pt A):51-6. doi: 10.1016/j.heares.2015.07.014. Epub 2015 Aug 12. PMID 26276418
- [Background] Vasama JP, Linthicum FH Jr. Temporal bone histopathology case of the month: otosclerosis. Am J Otol. 1998 May;19(3):398-9. No abstract available. PMID 9596194
- [Background] Veillon F, Riehm S, Emachescu B, Haba D, Roedlich MN, Greget M, Tongio J. Imaging of the windows of the temporal bone. Semin Ultrasound CT MR. 2001 Jun;22(3):271-80. doi: 10.1016/s0887-2171(01)90011-3. PMID 11451100
- [Background] Chole RA, McKenna M. Pathophysiology of otosclerosis. Otol Neurotol. 2001 Mar;22(2):249-57. doi: 10.1097/00129492-200103000-00023. PMID 11300278
- [Background] Wegner I, van Waes AM, Bittermann AJ, Buitinck SH, Dekker CF, Kurk SA, Rados M, Grolman W. A Systematic Review of the Diagnostic Value of CT Imaging in Diagnosing Otosclerosis. Otol Neurotol. 2016 Jan;37(1):9-15. doi: 10.1097/MAO.0000000000000924. PMID 26649602
- [Background] Gros A, Vatovec J, Sereg-Bahar M. Histologic changes on stapedial footplate in otosclerosis. Correlations between histologic activity and clinical findings. Otol Neurotol. 2003 Jan;24(1):43-7. doi: 10.1097/00129492-200301000-00010. PMID 12544027
- [Background] Husain Q, Lin KF, Selesnick SH. Stapes prosthesis length and hearing outcomes. Laryngoscope. 2018 Mar;128(3):722-726. doi: 10.1002/lary.26700. Epub 2017 May 31. PMID 28561306
- [Background] Fayad JN, Semaan MT, Meier JC, House JW. Hearing results using the SMart piston prosthesis. Otol Neurotol. 2009 Dec;30(8):1122-7. doi: 10.1097/MAO.0b013e3181be645d. PMID 19816231
- [Background] Avan P, Giraudet F, Buki B. Importance of binaural hearing. Audiol Neurootol. 2015;20 Suppl 1:3-6. doi: 10.1159/000380741. Epub 2015 May 19. PMID 25998698
- [Background] Weiss R, Leinung M, Baumann U, Weissgerber T, Rader T, Stover T. Improvement of speech perception in quiet and in noise without decreasing localization abilities with the bone conduction device Bonebridge. Eur Arch Otorhinolaryngol. 2017 May;274(5):2107-2115. doi: 10.1007/s00405-016-4434-2. Epub 2016 Dec 28. PMID 28032241
- [Background] Gartrell BC, Jones HG, Kan A, Buhr-Lawler M, Gubbels SP, Litovsky RY. Investigating long-term effects of cochlear implantation in single-sided deafness: a best practice model for longitudinal assessment of spatial hearing abilities and tinnitus handicap. Otol Neurotol. 2014 Oct;35(9):1525-32. doi: 10.1097/MAO.0000000000000437. PMID 25158615
- [Background] Schleich P, Nopp P, D'Haese P. Head shadow, squelch, and summation effects in bilateral users of the MED-EL COMBI 40/40+ cochlear implant. Ear Hear. 2004 Jun;25(3):197-204. doi: 10.1097/01.aud.0000130792.43315.97. PMID 15179111
- [Background] Jansen S, Luts H, Wagener KC, Kollmeier B, Del Rio M, Dauman R, James C, Fraysse B, Vormes E, Frachet B, Wouters J, van Wieringen A. Comparison of three types of French speech-in-noise tests: a multi-center study. Int J Audiol. 2012 Mar;51(3):164-73. doi: 10.3109/14992027.2011.633568. Epub 2011 Nov 28. PMID 22122354
- [Background] De Seta E, Rispoli G, Balsamo G, Covelli E, De Seta D, Filipo R. Indication for surgery in otosclerotic patients with unilateral hearing loss. Otol Neurotol. 2009 Dec;30(8):1116-21. doi: 10.1097/MAO.0b013e3181bc3c22. PMID 19752765
- [Derived] Baguant A, Schmerber S, Baguant K, Quatre R. Binaural squelch effect in unilateral otosclerosis surgery: comparison of speech intelligibility in noise before-after surgery. Eur Arch Otorhinolaryngol. 2022 Mar;279(3):1301-1310. doi: 10.1007/s00405-021-06797-3. Epub 2021 Apr 12. PMID 33846850